CLINICAL TRIAL: NCT02865772
Title: Reference Ranges of Lamellar Body Counts on Gastric Aspirate in Healthy Term Newborns
Brief Title: Lamellar Body Counts on Gastric Aspirate in Healthy Term Newborns
Status: Completed | Type: Observational
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Sema Arayici, Principal Investigator, Zekai Tahir Burak Women's Health Research and Education Hospital
Other Study IDs: 14/2014
Record Dates: First submitted 2016-08-02; First posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Infant, Newborn, Diseases
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — gastric aspiration fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- observational: healthy newborns

SUMMARY:
The aim of this study to determine the reference ranges of LBC on gastric aspirate in healthy term newborns.

DETAILED DESCRIPTION:
Lamellar bodies represent the storage form of lung surfactant. Surfactant is produced in alveolar type II cells and transported to the alveolar surface as lamellar bodies. Lamellar bodies are present in the amniotic fluid and also gastric aspirate.It has become a preferred test for determine fetal lung maturity, because of the rapid, inexpensive, easily accessible and easily applicable method.

ELIGIBILITY:
Inclusion Criteria:

* infants born at ≥ 37 weeks of gestation and birth weight ≥ 2500 g

Exclusion Criteria:

* intubated immediately after birth, infants with respiratory distress, infants with gestational pathology that can influence fetal lung maturity (cases with premature rupture of membranes, preeclampsia/eclampsia, gestational diabetes, oligohydramnios/polyhidramnios or antenatal steroid use), infants with major congenital or chromosomal abnormalities and lack of parental consent, therapeutic infusion was given in the amniotic cavity or if gastric aspirate contaminated by meconium, pus or blood.

Ages: 10 Minutes to 30 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: healthy newborns
Sampling Method: Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
normal levels of lamellar body counts on gastric aspirate in healthy term newborns. | 2 months

IPD SHARING:
Plan to Share IPD: Undecided